CLINICAL TRIAL: NCT01273857
Title: Phase I Study of Cardiac Progenitor Cell Therapy in Patients With Single Ventricle Physiology
Brief Title: Transcoronary Infusion of Cardiac Progenitor Cells in Patients With Single Ventricle Physiology
Acronym: TICAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Okayama University (Other)
Collaborators: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Principal Investigator, Hidemasa Oh, MD, MD., Ph.D., Okayama University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MHLW10103228
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Hypoplastic Left Heart Syndrome; Single Ventricle; Heart Failure
Keywords: Cardiac progenitor cells; Cell therapy; Hypoplastic Left Heart Syndrome; Single Ventricle; Norwood; Sano modification; Glenn; Fontan
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Univentricular Heart; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator): Subjects will undergo standard staged-procedures without cell infusion
  Interventions: Procedure: staged shunt procedure
- Cell infusion (Experimental): Subjects will receive transcoronary infusion of autologous cardiosphere-derived cells 1 month after staged shunt procedure
  Interventions: Procedure: Autologous cardiac progenitor cell transplantation; Procedure: staged shunt procedure

INTERVENTIONS:
Procedure: Autologous cardiac progenitor cell transplantation — Patients will receive 0.3 million / kg of autologous cardiac progenitor cells via intracoronary delivery 1 month after cardiac surgery. Follow-up visits 3 months to 1 year after cell injection will need to prospectively verify the clinical, laboratory, and safety-related data.
  Other Names: Cardiosphere-derived cells
  Arms: Cell infusion
Procedure: staged shunt procedure — Norwood-Glenn, Glenn, or Fontan procedure will be applied

SUMMARY:
Hypoplastic left heart syndrome (HLHS) and related anomalies involved a single ventricle are characterized by hypoplasia of the left heart and the aorta with compromised systemic cardiac output. Infants with the syndrome generally undergo a staged surgical approach in view of an ultimate Fontan procedure. Although long-term survival in patients with HLHS and related single ventricle physiology has improved markedly with advances in medical and surgical therapies, a growing number of infants will ultimately require heart transplantation for end-stage heart failure due to several potential disadvantages include a negative effect on right ventricular function, arrhythmia, additional volume load via regurgitation from the nonvalved shunt, and impaired growth of the pulmonary artery.

Risk factors for poor outcome of heart transplantation with HLHS and single ventricle physiology are older age at transplantation and previous Fontan operation. New strategies are needed to improve the underlying transplant risks proper for the Fontan failure patients.

Emerging evidence suggests that heart-derived stem/progenitor cells can be used to improved cardiac function in patients with ischemic heart disease. In this trial, the investigators aimed to test the safety and feasibility of intracoronary injection of autologous cardiac progenitor cells in patients with HLHS and related single ventricle anomalies and that could improve ventricular function at 3 months' follow up.

DETAILED DESCRIPTION:
Autologous cardiac progenitor cells are isolated from patients' own cardiac tissues obtained during palliative shunt procedure. Patients will receive 0.3 million/kg of autologous cardiac progenitor cells via intracoronary delivery 1 month after cardiac surgery. Follow-up visits 3 months to 1 year after cell injection will need to prospectively verify the clinical, laboratory, and safety-related data.

ELIGIBILITY:
Inclusion Criteria:

* Infants with hypoplastic left heart syndrome and related single ventricle anomalies undergoing first to third palliative shunt surgeries will be recruited into the study.
* Patients between 0 and 6 years of age are eligible if written informed consent can be obtained.

Exclusion Criteria:

* Cardiogenic shock
* Eisenmenger syndrome
* Uncontrollable arrhythmia
* Severe chronic diseases
* Infections
* Cancer
* Unwillingness to participate

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hidemasa Oh, M.D., Ph.D., Principal Investigator — Department of Regenerative Medicine, Center for Innovative Clinical Medicine, Okayama University Hospital
Locations (1):
- Department of Regenerative Medicine, Center for Innovative Clinical Medicine, Okayama University Hospital, Okayama, Japan

REFERENCES:
- [Background] Takehara N, Tsutsumi Y, Tateishi K, Ogata T, Tanaka H, Ueyama T, Takahashi T, Takamatsu T, Fukushima M, Komeda M, Yamagishi M, Yaku H, Tabata Y, Matsubara H, Oh H. Controlled delivery of basic fibroblast growth factor promotes human cardiosphere-derived cell engraftment to enhance cardiac repair for chronic myocardial infarction. J Am Coll Cardiol. 2008 Dec 2;52(23):1858-1865. doi: 10.1016/j.jacc.2008.06.052. PMID 19038683
- [Background] Tateishi K, Takehara N, Matsubara H, Oh H. Stemming heart failure with cardiac- or reprogrammed-stem cells. J Cell Mol Med. 2008 Dec;12(6A):2217-32. doi: 10.1111/j.1582-4934.2008.00487.x. Epub 2008 Aug 27. PMID 18754813
- [Background] Tateishi K, Ashihara E, Takehara N, Nomura T, Honsho S, Nakagami T, Morikawa S, Takahashi T, Ueyama T, Matsubara H, Oh H. Clonally amplified cardiac stem cells are regulated by Sca-1 signaling for efficient cardiovascular regeneration. J Cell Sci. 2007 May 15;120(Pt 10):1791-800. doi: 10.1242/jcs.006122. PMID 17502484
- [Background] Tateishi K, Ashihara E, Honsho S, Takehara N, Nomura T, Takahashi T, Ueyama T, Yamagishi M, Yaku H, Matsubara H, Oh H. Human cardiac stem cells exhibit mesenchymal features and are maintained through Akt/GSK-3beta signaling. Biochem Biophys Res Commun. 2007 Jan 19;352(3):635-41. doi: 10.1016/j.bbrc.2006.11.096. Epub 2006 Nov 27. PMID 17150190
- [Result] Ishigami S, Ohtsuki S, Tarui S, Ousaka D, Eitoku T, Kondo M, Okuyama M, Kobayashi J, Baba K, Arai S, Kawabata T, Yoshizumi K, Tateishi A, Kuroko Y, Iwasaki T, Sato S, Kasahara S, Sano S, Oh H. Intracoronary autologous cardiac progenitor cell transfer in patients with hypoplastic left heart syndrome: the TICAP prospective phase 1 controlled trial. Circ Res. 2015 Feb 13;116(4):653-64. doi: 10.1161/CIRCRESAHA.116.304671. Epub 2014 Nov 17. PMID 25403163
- [Derived] Hirai K, Sawada R, Hayashi T, Araki T, Nakagawa N, Kondo M, Yasuda K, Hirata T, Sato T, Nakatsuka Y, Yoshida M, Kasahara S, Baba K, Oh H; TICAP/PERSEUS Study Group. Eight-Year Outcomes of Cardiosphere-Derived Cells in Single Ventricle Congenital Heart Disease. J Am Heart Assoc. 2024 Nov 19;13(22):e038137. doi: 10.1161/JAHA.124.038137. Epub 2024 Nov 11. PMID 39526355
- [Derived] Sano T, Ousaka D, Goto T, Ishigami S, Hirai K, Kasahara S, Ohtsuki S, Sano S, Oh H. Impact of Cardiac Progenitor Cells on Heart Failure and Survival in Single Ventricle Congenital Heart Disease. Circ Res. 2018 Mar 30;122(7):994-1005. doi: 10.1161/CIRCRESAHA.117.312311. Epub 2018 Jan 24. PMID 29367212
- [Derived] Tarui S, Ishigami S, Ousaka D, Kasahara S, Ohtsuki S, Sano S, Oh H. Transcoronary infusion of cardiac progenitor cells in hypoplastic left heart syndrome: Three-year follow-up of the Transcoronary Infusion of Cardiac Progenitor Cells in Patients With Single-Ventricle Physiology (TICAP) trial. J Thorac Cardiovasc Surg. 2015 Nov;150(5):1198-1207, 1208.e1-2. doi: 10.1016/j.jtcvs.2015.06.076. Epub 2015 Jul 8. PMID 26232942

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Cell Infusion
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Cell Infusion | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.5 (1.7) | 2.1 (1.2) | 1.7 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  Japan | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Evaluation and Major Cardiac Adverse Events Related to Transcoronary Infusion of Cardiac Progenitor Cells
Description: Feasibility was assessed by number of participants discontinued the study due to adverse events or number of participants received unsuccessful cell delivery by study physician. Unsuccessful was defined as failure of coronary selection of guiding catheter or direct cell infusion.
  The primary end point is to monitor major adverse cardiac events include death, sustained/symptomatic ventricular tachycardia, aggravation of heart failure, new myocardial infarction, unplanned cardiovascular operation for cardiac tamponade and infection in the first month after injection, and serially afterwards.
Time Frame: 3 months to 1 year after cell transplantation
Measure: Number; unit: participants
Arm/Group | Control | Cell Infusion
Number analyzed (Participants) | 7 | 7
participants | 0 | 0

2. Secondary Outcome: Serious Adverse Events
Description: The incidence of hospitalization for heart failure, ventricular arrhythmia, general infection, and renal and hepatic dysfunction by CDC treatment.
Time Frame: 3 months to 1 year after cell transplantation
Measure: Number; unit: participants
Arm/Group | Control | Cell Infusion
Number analyzed (Participants) | 7 | 7
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 years
Arm/Group | Control | Cell Infusion
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No